CLINICAL TRIAL: NCT06953440
Title: The Effect of Dexamethasone Submucosal Injection After Third Molar Surgery on Trismus and Edema
Brief Title: The Effect of Dexamethasone Submucosal Injection After Surgical Extraction of Lower Impacted Third Molars on Trismus and Edema
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Lojain Bassyoni, Oral and Maxillofacial Surgery Consultant and Assistant Professor, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 225-11-23
Record Dates: First submitted 2025-02-11; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Swelling/ Edema; Trismus
Keywords: Extraction; third molar; wisdom teeth; dexamethasone; steroids; submucosal
MeSH Terms: conditions — Edema; Trismus | interventions — dexamethasone 21-phosphate; Saline Solution

STUDY DESIGN:
Intervention Model Description: There will be two groups. The test group will receive 4mg/1ml dexamethasone submucosal injection at the buccal vestibule next to the surgical site. The control group will receive 1 ml of normal saline injection in the buccal vestibule next to the surgical site.
  The primary objective of this study is to compare mean change in trismus and mean edema between 2 independent groups.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: To ensure that the patient and OMFS resident were blinded in this study, the corticosteroid and placebo injections were of the same color and size, were stored in similar syringes, and were coded as drug 1 or drug 2. The OMFS resident received the syringe corresponding to the patient's random allocation prior to the beginning of the procedure. The number of the drug was recorded in the patient file. Then, the drug was administered in the buccal vestibule next to the site of extraction after surgery. Thus, the patient, surgeon, and the person responsible for the assessments of swelling and trismus were masked to the type of medication used during each surgical procedure. The drugs used in the different surgeries were only revealed after the acquisition and analysis of all data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexamethasone Group (Experimental): Patient received 4 milligrams of dexamethasone
  Interventions: Drug: Dexamethasone Sodium Phosphate Injection
- Control Group (Placebo Comparator): Patient received 4 milligrams of normal saline solution
  Interventions: Other: Normal Saline (Placebo)

INTERVENTIONS:
Drug: Dexamethasone Sodium Phosphate Injection — Patients will receive 4 milligrams of dexamethasone submucosal injection next to the extraction site.
  Arms: Dexamethasone Group
Other: Normal Saline (Placebo) — Patients will receive 4 milligrams of normal saline solution next to the extraction site.
  Arms: Control Group

SUMMARY:
This clinical trial aims to investigate whether dexamethasone decreases edema and trismus in adults undergoing lower third molar surgical extraction.

The main question it aims to answer is:

Does dexamethasone submucosal injection have a positive impact on trismus and edema after third molar surgery compared to conventional postoperative prescription?

Participants will:

* Be administered with dexamethasone submucosal injection or a placebo after the surgery.
* Visit the clinic three times the week after the extraction for follow-up.

DETAILED DESCRIPTION:
Patients will be randomly allocated to the test group or the control group by an allocation sequence that is done by the statistician.

To ensure that the patient and OMFS resident are blinded in this study, the corticosteroid and placebo injections are of the same color and size, are stored in similar bottles, and are coded as drug 1 or drug 2. Additionally, they will be placed in sealed envelopes by a dental assistant.

The OMFS resident will withdraw an envelope randomly. The number is recorded in the patient file. Then, the drug will be administered in the buccal vestibule next to the site of extraction after surgery. Thus, the patient, surgeon, and the person responsible for the assessments of swelling and trismus are masked to the type of medication used during each surgical procedure. The drugs used in the different surgeries are only revealed after the acquisition and analysis of all data. Baseline and follow-up measurements will be measured by a standardized ruler. At the first visit, interincisal distance will be recorded to measure trismus. Distance from the angle of the mandible to the outer canthus of the eye, distance from the tragus of the ear to the corner of the mouth, and distance from the tragus of the ear to soft tissue pogonion will be recorded and their mean will be calculated to measure edema. Pell and Gregory classification of the tooth and impaction angulation will be recorded. Facial symmetry and whether the angle of the mandible is palpable or not will be recorded as well. The number of drug that was given to the patient will be recorded.

At the 2nd, 4th, and 7th visits, interincisal distance will be recorded to measure trismus. Distance from the angle of the mandible to the outer canthus of the eye, distance from the tragus of the ear to the corner of the mouth, and distance from the tragus of the ear to soft tissue pogonion will be recorded to measure edema. Facial symmetry and whether the angle of the mandible is palpable or not will be recorded. Whether the patient is able to interact socially or not. If not, was it due to edema, feeling sick, or bad mood. The patient's ability to work, the patient's ability to eat the food he is used to eating, and the presence of sleep impairment will be recorded as well.

Surgery will be done by calibrated OMFS residents. After the surgery, the surgeon will use the preassigned randomly picked envelope and administer it in the buccal vestibule next to the surgical site. Patients will be followed up in the 2nd, 4th, and 7th postoperative days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with impacted lower third molars requiring surgical extraction.
* Adults over the age of 18 years old.
* American Society of Anaesthesiologists (ASA) 1, and ASA 2

Exclusion Criteria:

* Patients with preoperative intraoral or extraoral swelling.
* Patients requiring simple extraction (Class I group A according to Pell and ---Gregory classification).
* Patients with uncontrolled systemic disease such as uncontrolled diabetic - patients.
* Patients who are allergic to corticosteroids.
* Patients who are contraindicated to use corticosteroids such as uncontrolled diabetic patients, and osteoporotic patients.
* Patients who require extraction of additional teeth at the same visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Trismus and Swelling | From the day of extraction, the 2nd day of surgery, 4th day, and 7th day of surgery.
  Baseline and follow-up measurements will be measured by a standardized ruler. At the first visit, interincisal distance will be recorded in millimeters to measure trismus. Distance from the angle of the mandible to the outer canthus of the eye, distance from the tragus of the ear to the corner of the mouth, and distance from the tragus of the ear to soft tissue pogonion will be recorded in millimeters and their mean will be calculated to measure edema. Pell and Gregory classification of the tooth and impaction angulation will be recorded. Facial symmetry and whether the angle of the mandible is palpable or not will be recorded as well.
  At the 2nd, 4th, and 7th visits, interincisal distance will be recorded in millimeters to measure trismus. Distance from the angle of the mandible to the outer canthus of the eye, distance from the tragus of the ear to the corner of the mouth, and distance from the tragus of the ear to soft tissue pogonion will be recorded in millimeters

SECONDARY OUTCOMES:
Social Interaction | Patients will be followed up in the 2nd, 4th, and 7th postoperative days.
  Whether the patient is able to interact socially or not, if not, was it due to edema, feeling sick, or bad mood.
  The patient will be asked a yes or no question, and their answer will be recorded.
Work Ability | Patients will be followed up in the 2nd, 4th, and 7th postoperative days.
  Whether the patient is able to work on his job or perform daily chores.
  The patient will be asked a yes or no question, and their answer will be recorded.
Eating Ability | Patients will be followed up in the 2nd, 4th, and 7th postoperative days.
  Whether the patient can eat the food he is used to.
  The patient will be asked a yes or no question, and their answer will be recorded.
Sleep Impairment | Patients will be followed up in the 2nd, 4th, and 7th postoperative days.
  Whether the patient is able to sleep without impairment.
  The patient will be asked a yes or no question, and their answer will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- King Abdulaziz University, Faculty of Dentistry, Jeddah, Mecca Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
All data gathered and agreed upon by the institution's research ethical committee throughout the conduction of the clinical trial will be shared at the time of publication.

REFERENCES:
- [Background] Hou C, Liu F, Liu C. Comparison of Submucosal With Intramuscular or Intravenous Administration of Dexamethasone for Third Molar Surgeries: A Systematic Review and Meta-Analysis. Front Surg. 2021 Aug 10;8:714950. doi: 10.3389/fsurg.2021.714950. eCollection 2021. PMID 34447785
- [Background] Grossi GB, Maiorana C, Garramone RA, Borgonovo A, Beretta M, Farronato D, Santoro F. Effect of submucosal injection of dexamethasone on postoperative discomfort after third molar surgery: a prospective study. J Oral Maxillofac Surg. 2007 Nov;65(11):2218-26. doi: 10.1016/j.joms.2006.11.036. PMID 17954317
- [Background] Wanithanont P, Chaiyasamut T, Vongsavan K, Bhattarai BP, Pairuchvej V, Kiattavorncharoen S, Wongsirichat N. Comparative efficiency of the preoperative pterygomandibular space injection of two doses of dexamethasone in mandibular third molar surgery. J Dent Anesth Pain Med. 2021 Feb;21(1):29-39. doi: 10.17245/jdapm.2021.21.1.29. Epub 2021 Jan 29. PMID 33585682
- [Background] Warraich R, Faisal M, Rana M, Shaheen A, Gellrich NC, Rana M. Evaluation of postoperative discomfort following third molar surgery using submucosal dexamethasone - a randomized observer blind prospective study. Oral Surg Oral Med Oral Pathol Oral Radiol. 2013 Jul;116(1):16-22. doi: 10.1016/j.oooo.2012.12.007. Epub 2013 Feb 28. PMID 23453611
- [Background] Mojsa IM, Pokrowiecki R, Lipczynski K, Czerwonka D, Szczeklik K, Zaleska M. Effect of submucosal dexamethasone injection on postoperative pain, oedema, and trismus following mandibular third molar surgery: a prospective, randomized, double-blind clinical trial. Int J Oral Maxillofac Surg. 2017 Apr;46(4):524-530. doi: 10.1016/j.ijom.2016.11.006. Epub 2016 Dec 21. PMID 28012633
- [Background] Parhizkar P, Schmidlin PR, Bornstein MM, Fakheran O. Can adjunctive corticosteroid therapy improve patient-centered outcomes following third molar surgery? A systematic review. Med Oral Patol Oral Cir Bucal. 2022 Sep 1;27(5):e410-e418. doi: 10.4317/medoral.25177. PMID 35975802
- [Background] Moraschini V, Hidalgo R, Porto Barboza Ed. Effect of submucosal injection of dexamethasone after third molar surgery: a meta-analysis of randomized controlled trials. Int J Oral Maxillofac Surg. 2016 Feb;45(2):232-40. doi: 10.1016/j.ijom.2015.09.008. Epub 2015 Oct 14. PMID 26458538
- [Background] Kiencalo A, Jamka-Kasprzyk M, Panas M, Wyszynska-Pawelec G. Analysis of complications after the removal of 339 third molars. Dent Med Probl. 2021 Jan-Mar;58(1):75-80. doi: 10.17219/dmp/127028. PMID 33789003
- [Background] Aljafar A, Alibrahim H, Alahmed A, AbuAli A, Nazir M, Alakel A, Almas K. Reasons for Permanent Teeth Extractions and Related Factors among Adult Patients in the Eastern Province of Saudi Arabia. ScientificWorldJournal. 2021 Feb 22;2021:5534455. doi: 10.1155/2021/5534455. eCollection 2021. PMID 33688305
- See also: Google drive link that contains all information regarding the study — https://drive.google.com/drive/folders/1LIwA4RHf660gjAvCJ0mFQ3bTMZx0FlDA?usp=drive_link